CLINICAL TRIAL: NCT02267590
Title: Clinical Validation of Biomarkers Determining Resistance to BTK Inhibition With Ibrutinib in Mantle Cell Lymphoma & Chronic Lymphocytic Leukaemia - Stage 1
Brief Title: Tissue Collection for Biomarkers Determining Resistance to Ibrutinib
Acronym: CLARITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: University Hospital Plymouth NHS Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4187
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Mantle Cell Lymphoma; Chronic Lymphocytic Leukaemia
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Leukemia, B-Cell

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20mls of PB in EDTA; 5ml of BM in EDTA and/or tissue biopsy (fresh/frozen/FFPE) and/or pleural/ascitic fluid containing tumour cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MCL: 80-100 samples from 60- 70 patients: Mantle Cell lymphoma patients
- CLL: 15-20 samples from 10-15 patients: Chronic lymphocytic leukaemia patients

SUMMARY:
Clinical validation of biomarkers determining resistance to BTK inhibition with Ibrutinib in Mantle Cell Lymphoma and Chronic Lymphocytic Leukaemia Stage 1.

DETAILED DESCRIPTION:
With the recent FDA approval of Ibrutinib for the management of relapsed/refractory MCL and CLL, we are entering an exciting phase in the management of these conditions. A crucial next step is to validate biomarkers that predict clinical activity of Ibrutinib in order to tailor therapy and maximise benefit to patients. The recently opened named patient supply (NPS) of ibrutinib in the UK provides an excellent window of opportunity for these studies.

The investigators have set up a collaboration with Professor Simon Rule (Plymouth) and Dr George Follows (Cambridge), who are carrying out a prospective data collection study for patients entered on to the NPS. With the help of our collaborators the investigators will be able to identify centres in the NHS for collection of samples. Patients entered on to the NPS will be provided an information sheet and research specific consent form following which samples from consenting patients will be transferred to the Royal Marsden Hospital (RMH) for storage. Samples will be logged and tracked using a secure database. Samples for research will be collected at the same time as routine sampling and therefore no additional sampling will be required. For each patient, consent will be obtained for pretreatment, progression as well as any diagnostic samples taken or stored and patients will require to be on the study for at least 24 months from the start of their treatment. The collection will end 24 months after the last patient commences treatment on the NPS.

Once we have an idea of the number of patient samples we can collect, the second stage of this study will be initiated and will involve molecular screening of samples at RMH for biomarkers of resistance. The data from the molecular studies will then be correlated with the clinical response data from our collaborators for clinical validation.

ELIGIBILITY:
Inclusion Criteria:

* All patients entered into the Ibrutinib NPS for relapsed refractory MCL and CLL in the UK and who consent to have biological material stored for this research will be included in the study. Patients who have already commenced treatment with Ibrutinib will also be eligible whether or not they are responding.

Exclusion Criteria:

* All samples received will undergo histological (or morphological) review and immunophenotyping. The following samples will be excluded-

  1. Samples not satisfying the criteria for diagnosis of CLL or MCL.
  2. Samples with evidence of high grade transformation (e.g. Richter's transformation of CLL).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Ibrutinib named patient supply (NPS) was introduced across the NHS for relapsed/ refractory CLL in April this year. Patients with relapsed/ refractory MCL were allowed to enter this programme in September. The NPS for CLL is likely to be open until the 30th of September this year while MCL patients can access Ibrutinib until the end of November. Strict inclusion and exclusion criteria have been set out for the NPS and patients are required to be screened through an online portal prior to entry on to the programme. The NPS provides an excellent window of opportunity to collect patient samples for this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Total number of MCL and CLL patient samples collected, both pre-treatment and at progression. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom